CLINICAL TRIAL: NCT06688370
Title: The Performance and Safety of Petit Drill in the French Paediatric Population: a Post-market Clinical Follow-up.
Brief Title: The Performance and Safety of Petit Drill in the French Paediatric Population: a Post-market Clinical Follow-up Study
Acronym: Touxpetit
Status: Terminated | Type: Observational
Why Stopped: Due to difficulty in recruiting patients, the Sponsor decided to prematurely stop the study
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: CEN Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS17379; 2023-A01929-36 (Registry Identifier: ANSM)
Record Dates: First submitted 2024-03-15; First posted 2024-11-14 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sore-throat; Cough
Keywords: dry cough; Petit Drill; throat irritation; sore throat
MeSH Terms: conditions — Pharyngitis; Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Petit Drill: Participants who received treatment with the syrup (at least once) as long as necessary from D1 to D3, according to parent's judgement.
  Interventions: Device: Petit Drill

INTERVENTIONS:
Device: Petit Drill — Day 1: 2-4 doses, including one of the daily doses taken at bedtime. Days 2 and 3: 3 to 4 doses, including one of the daily doses taken at bedtime.

SUMMARY:
Demulcent or soothing substance is the currently recommended option to alleviate throat irritation associated to cough and sore throat in children under 6 years. The intended benefit to the patient of Petit Drill is to calm throat irritation (sore throat) associated to dry cough in infants starting at 6 months of age and in children up to 6 years of age. This intended benefit sustained by the properties of the formula is recognized and promoted by the World Health Organization, health authorities and current textbooks to have a positive impact on patient management for the targeted population (infant / child).

This study aimed at assessing the performance of the syrup in real-life context, in children presenting throat irritation associated with dry cough to support the conclusion of clinical evaluation report.

DETAILED DESCRIPTION:
Pediatric patients were recruited by pharmacist in community settings, who briefly presented the clinical investigation to the parent who purchases Petit Drill for his/her child.

The pharmacist provided the interested parent with the study information note and transferred the parent's name and contact details to the clinical investigation centre. The parent was then contacted to take part in the remote inclusion visit with a site investigator, scheduled on the same day of Petit Drill delivery. During the inclusion visit, once consent has been signed, the investigator verified eligibility criteria, and collected baseline data.

The follow-up periods lasted as long as the child received the syrup, but it should not exceed 3 days and 3 nights. The parent completed daily questionnaires and recorded the child's syrup intake in a secure mobile application designed for patient reported outcomes (PROs).

Of note, due to the premature discontinuation of the study, all statistical analyses initially planned in the Statistical Analysis Plan (SAP) were not conducted. All study outcomes were analyzed using descriptive statistics. Therefore, results presented hereafter are limited to few study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls, 6 months to 6 years of age;
* With one of his/her parents/legal guardian purchases Petit Drill in a participating pharmacy in accordance with recommendations for use (regarding age and type of cough);
* For infants between 6 months and 12 months of age - a confirmed prescription from a treating physician;
* With an acute dry cough lasting less than 48 hours
* With a score ≥ 3 at least for 3 of the 5 items of PCQ, (based on assessment of the night before inclusion);
* For whom child-minding will allow to respect the recommended daily doses of Petit Drill during the 3 day-treatment;
* With a parent/legal guardian having a smartphone allowing using the ePRO App. NursTrial®;
* With a parent/legal guardian able to understand and to complete to the questionnaires in timely manner;
* With parent(s)/legal guardian who provide their signed informed consent for the child's enrolment in the study.

Exclusion Criteria:

* Presenting with one of the following conditions: Chronic respiratory illness such as asthma, recurrent wheezing associated to viral infections and bronchitis or lower respiratory infections, such as bronchitis, bronchiolitis, and pneumonia or angina, otitis, or sinusitis or persistent cough lasting more than 3 weeks, whatever the etiology or gastrointestinal pathology, involving vomiting, nausea, or diarrhoea.
* With ongoing use of paracetamol, and/or homeopathic products against cough.
* Having had corticosteroid treatment, antibiotics, antihistaminic or any cough medication (such as, but not limited to, Phytoxil, Arkotoux) in the previous 15 days since inclusion.
* With a brother/sister already included in the present clinical investigation (If several children are eligible in the same household, only one will be enrolled at random).
* Enrolled in another clinical trial or being in a period of exclusion from a previous clinical trial.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric population presented with acute dry cough
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT ALQUIER, Principal Investigator — Pharmacist; GUY DUTAU, Study Chair — pediatrician pulmologist
Locations (1):
- Cen Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Petit Drill: Participants who received treatment with the syrup (at least once) as long as necessary from D1 to D3, according to parent's judgement.
  Petit Drill: Day 1: 2-4 doses, including one of the daily doses taken at bedtime.
  Days 2 and 3: 3 to 4 doses, including one of the daily doses taken at bedtime.
Period: Overall Study
Arm/Group | Petit Drill
Started | 12
Completed (Completed refers to the completion of the Performance Analysis Set) | 7
Not Completed | 5
Not completed — Discontinued the treatment | 1
Not completed — Prohibited treatment taken | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population: the analysis population consists of patients who were included in this clinical investigation after fulfilling all eligibility criteria.
Arm/Group | Petit Drill
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: year] | 3.1 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Rank of sibling [Count of Participants; unit: Participants]
  Single child | 3
  First | 4
  Second | 2
  Third | 2
  Fourth | 1
Description of study population (home region) [Count of Participants; unit: Participants]
  Bourgogne Franche-Comté | 1
  Centre-Val de Loire | 1
  Grand Est | 3
  Hauts-de-France | 2
  Nouvelle-Aquitaine | 3
  Occitanie | 2

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Pediatric Cough Questionnaire (PCQ) Total Score - Percentage of Children With a 3-point Decrease From Baseline After up to 3-day Treatment With Petit Drill
Description: Percentage of children with a 3 point-decrease (minimal clinical significance) of the Pediatric Cough Questionnaire (PCQ) total score from baseline after up to 3 day-treatment with Petit Drill.
  PCQ refers to a past night recall of 5 questions, each scored from 0 "Not at all" to 5 "Extremely" using a 6-point Likert scale.
  PCQ Total score consists of the sum of each score and ranges from 0 to 25.
Time Frame: up to 3 days
Population: Performance population which consists of all patients from the safety population without any major deviation from the protocol and for whom at least one evaluation of the primary outcome is available after treatment initiation (baseline and last assessment) and whose parent(s) or legal guardian did not withdraw their consent at any time.
  Due to the premature study discontinuation, analysis initially planned was not done, and all study outcomes were analyzed using descriptive statistics.
Measure: Count of Participants; unit: Participants
Arm/Group | Petit Drill
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Petit Drill Adherence
Description: Average number of times Petit Drill is administered in each 24-hour period
Time Frame: Day 1, day 2 and day 3
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Petit Drill
Number analyzed (Participants) | 12
Participants
  At least 1 day with 3 doses | 6
  1 day with 4 doses | 1
  less than 3 doses received at all days | 5

3. Secondary Outcome: Parent's Satisfaction With Petit Drill
Description: Satisfaction is assessed using a study specific questionnaire. Responses measured using Likert scales. Not validated Questionnaire; 6 questions with different way to answers.
  Of note, parents were not considered enrolled but did contribute to this assessment.
Time Frame: Day 3
Population: Full Analysis Set (FAS) population: the analysis population consists of patients who were included in this clinical investigation after fulfilling all eligibility criteria. Of note, parents were not considered enrolled but did contribute to this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Petit Drill
Number analyzed (Participants) | 9
Participants
  Quality of therapeutic management: excellent | 2
  Quality of therapeutic management: good | 5
  Quality of therapeutic management: fair | 1
  Quality of therapeutic management: poor | 1
  Response to the child's needs: almost all were met | 2
  Response to the child's needs: most were met | 4
  Response to the child's needs: only few were met | 3
  Response to the child's needs: none were met | 0
  Willingness to recommend the syrup: yes generally | 2
  Willingness to recommend the syrup: yes definitely | 5
  Willingness to recommend the syrup: no | 2
  Satisfaction with information from Instruction For Use (IFU) to use treatment: quite dissatisfied | 0
  Satisfaction with information from IFU to use treatment: indifferent or mildly dissatisfied | 0
  Satisfaction with information from IFU to use treatment: mostly satisfied | 6
  Satisfaction with information from IFU to use treatment: very satisfied | 3
  Ease of syrup use: yes generally | 2
  Ease of syrup use: yes definitely | 7
  Ease of syrup use: no | 0
  Feeling that the child enjoyed the syrup taste: yes generally | 2
  Feeling that the child enjoyed the syrup taste: yes definitely | 7
  Feeling that the child enjoyed the syrup taste: no | 0

4. Secondary Outcome: Petit Drill Safety
Description: Number of participants with adverse events and adverse device effects coded by using the System Organ Class (SOC) and Preferred Term (PT) of the version 24.1 of the Medical Dictionary for Regulatory Activities (MedDRA) dictionary.
Time Frame: 3 days
Population: Safety population: the safety population will include all patients from the FAS population who used Petit Drill at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Petit Drill
Number analyzed (Participants) | 12
Participants
  Adverse events | 4
  Serious adverse events | 0
  Adverse device effect related to procedures | 1
  Adverse device effect related to device deficiency | 1
  Adverse event leading to permanent discontinuation | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected over days D1, D2, D3, D4
Groups:
- Petit Drill: Treatment with the syrup for as long as necessary from D1 to D3, according to parent's judgement.
  Petit Drill: Day 1: 2-4 doses, including one of the daily doses taken at bedtime.
  Days 2 and 3: 3 to 4 doses, including one of the daily doses taken at bedtime.
Arm/Group | Petit Drill
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Petit Drill (N=12)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 — This is an adverse device effect
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Tonsilitis (Respiratory, thoracic and mediastinal disorders) | 1
Underdose (Injury, poisoning and procedural complications) | 1 — This is an adverse device effect
Device use error (Injury, poisoning and procedural complications) | 1 — This is an adverse device effect
Vomiting (Gastrointestinal disorders) | 1 — This is an adverse device effect
Fatigue (General disorders) | 1

LIMITATIONS AND CAVEATS:
The main limitation of this study is the very small number of patients included and analyzed (12 patients in the safety analysis; 7 in performance), because the study had been stopped prematurely due to major recruitment difficulties.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT06688370/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT06688370/SAP_001.pdf